CLINICAL TRIAL: NCT04947423
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of the Efficacy and Safety of DPI-386 Nasal Gel for the Prevention of Nausea and Vomiting Associated With Motion
Brief Title: Nasal Gel for the Prevention of Nausea and Vomiting Associated With Motion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repurposed Therapeutics, Inc. (Industry)
Collaborators: Defender Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPI-386-MS-29
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness | interventions — Scopolamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DPI-386 Nasal Gel (Experimental): Each 0.12 gram of the gel contains 0.2 mg of scopolamine HBr
  Interventions: Drug: DPI-386 Nasal Gel
- Placebo (Placebo Comparator): Placebo Nasal Gel (0.12 g)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DPI-386 Nasal Gel — Subjects will self-administer DPI-386 Nasal Gel or Placebo
  Other Names: scopolamine
  Arms: DPI-386 Nasal Gel
Drug: Placebo — Subjects will self-administer DPI-386 Nasal Gel or Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 3, two-arm, randomized, double-blind, placebo-controlled, single dose efficacy and safety study evaluating the use of a nasal gel to prevent nausea and vomiting associated with motion

DETAILED DESCRIPTION:
Eligible participants will be randomized 1:1 to DPI-386 Nasal Gel or matching placebo nasal gel and assigned a time and date for travel on an ocean vessel. Participants will be asked to self-administer the study medication while the ship is in harbor. The Modified Performance Self-Assessment Questionnaire (mPSAQ) will be completed by each participant prior to the administration of nasal gel, approximately every 30 minutes of travel, and at the end of travel. The participants will complete the Nausea Assessment Scale (NAS) every 30 minutes afer dosing, and at the end of travel. The participants will also be asked to complete a Sopite Assessment Questionnaire (SAQ) and a Patient Global Assessment of Severity (PGI-S) at 4 hours to describe their travel experience. All questionnaires will be submitted for analysis. An exit interview will also be conducted.

The treatment phase will last approximately 4-5 hours

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written, informed consent prior to initiation of any study-related procedures, and ability in the opinion of the Investigator to understand and comply with all the requirements of the study, which includes abstaining from the use of prohibited medications.
2. Male and female participants, aged 18 to 70 years of age (inclusive);
3. Minimally susceptible to provocative motion as evidenced by at least two responses on the (MSSQ-short) of "Sometimes" or "Frequently";
4. Acceptable overall medical condition to be safely enrolled in and complete the study in the opinion of the Investigator;
5. Ability to take intranasal medication;
6. Males, non-fecund females (i.e., surgically sterilized, if procedure was done 6 months before screening or participant is 2 years postmenopausal), or females of childbearing potential using an acceptable method of birth control (i.e., condoms, diaphragm, spermicidal agents, cervical cap, copper intrauterine device, etc.) for a period of up to 30 days before dosing and for one month after dosing and must have a negative pregnancy test at screening;
7. Agree to adhere to the following lifestyle compliance considerations:

   1. Refrain from consumption of grapefruit and any substance containing grapefruit for 7 days prior to, during, and 7 days after study drug administration;
   2. Abstain from alcohol for 24 hours prior to the administration of study drug and through the ocean travel;
   3. Abstain from marijuana within the 7-day period prior to the Treatment Day and throughout Day 3..
8. Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) negative test, confirmed by Food and Drug Administration (FDA) authorized COVID-19 test < 7 days prior to study drug administration or no COVID 19 symptoms up to 10 days prior to study drug administration.

Exclusion Criteria:

Main Criteria for Exclusion:

1. Nauseated prior to boarding.
2. Mini-Mental State Examination score of <24;
3. Women of childbearing potential, or men whose sexual partner(s) is a woman of childbearing potential, who:

   1. Are or intend to become pregnant (including use of fertility drugs) during the study;
   2. Are nursing (female participants only);
   3. Are not using an acceptable, highly effective method of contraception until all follow-up procedures are complete.
4. Known allergic reactions to scopolamine or other anticholinergics;
5. Hospitalization or significant surgery requiring hospital admittance within the past 6 months;
6. Treatment with another investigational product within the past 30 days;
7. Donated blood or plasma or suffered significant blood loss within the past 30 days;
8. Chronic nausea caused by conditions such as irritable bowel syndrome, gastroparesis, cyclic vomiting syndrome or any other cause;
9. Having any of the following medical conditions within the last 2 years or if any of the following medical conditions were experienced more than 2 years ago and are deemed as clinically significant by the Investigator:

   1. Significant gastrointestinal disorder, asthma, or seizure disorders;
   2. History or current cardiovascular disease;
   3. History or current vestibular disorders;
   4. History or current narrow-angle glaucoma;
   5. History or current urinary retention problems;
   6. History or current alcohol or drug abuse;
   7. History or current nasal, nasal sinus or nasal mucosa surgery.
10. Currently taking any of the following medication types within the specified washout period:

    1. Any form of scopolamine (including Transderm Scop®/washout 5 days;
    2. Belladonna alkaloids/washout 14 days;
    3. Antihistamines (including meclizine/washout 14 days;
    4. Tricyclic antidepressants/washout 14 days;
    5. Muscle relaxants/washout 4 days, and;
    6. Nasal decongestants/washout 4 days.
11. Has used marijuana within the 7-day period prior to the Treatment Day. (Note: this criterion will only be confirmed at Eligibility Confirmation, not at Recruitment and Screening, although heavy users of marijuana can be determined ineligible at Screening. All potential study participants deemed eligible at Screening must be informed at that time that this requirement must be met at Eligibility Confirmation.)
12. Unwilling or unable to follow the medication restrictions or unwilling to wash-out the use of restricted medications as noted in Exclusion 10.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who report no vomiting within 4 hours after receiving study drug and no use of rescue treatment (e.g., dimenhydrinate) within 4 hours after receiving study drug (Complete Responders). | 4 hours
  Participants who report no vomiting within 4 hours after receiving study drug and no use of rescue treatment (e.g., dimenhydrinate) within 4 hours after receiving study drug

CONTACTS AND LOCATIONS:
Overall Officials: David Helton, Study Director — Defender Pharmaceuticals, Inc.
Locations (1):
- Santa Monica Clinical Trials, Santa Monica, California, United States